CLINICAL TRIAL: NCT06997354
Title: Validation of a Parental Questionnaire for Screening Children for Neurovisual Disorders
Status: Recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: QP-TNV
Record Dates: First submitted 2025-05-12; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Children Suffering From Cortical Visual Impairment
MeSH Terms: interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- questionnaire: Each parent has to complete a online questionnaire
  Interventions: Diagnostic Test: Questionnaire

INTERVENTIONS:
Diagnostic Test: Questionnaire — The parents have to complete a questionnaire

SUMMARY:
Some children present visual difficulties linked not to damage to the eye, but to damage to the brain. This type of dysfunction of the visual cerebral pathways leads, for example, to difficulties in recognition, visuomotor coordination or visuo-spatial disorders. These highly specific disorders are known as "cortical visual impairment" (CVI). Despite their real impact on children's development, these disorders are still poorly diagnosed in the French-speaking world. As a result, follow-up and care for these children are poorly adapted. A better understanding of neurovisual disorders and the availability of validated tools in French are therefore essential. Indeed, it is currently considered that 3 to 4% of children aged four to six, i.e. around one child per kindergarten class, have a CVI following a neuro-logical lesion acquired in the perinatal period.

Because of the lack of a valid tool in French, the aim of the present study is to provide the results of a validation study of a parental questionnaire for screening children with warning signs of CVI in French. This questionnaire will be offered online using the Qualtrics tool. In order to evaluate the relevance of this questionnaire, it will be proposed, on the one hand, to parents whose child (aged 3 to 12) does not present any particular developmental difficulties, and on the other hand, to parents whose child (aged 3 to 12) seems to present signs of neurovisual disorders. By comparing their answers, the investigators hope that certain questions will reveal elements typical of neurovisual disorders/CVI, thus demonstrating the relevance of this questionnaire in facilitating diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Parents of a child aged between 3 and 12
* Their mother tongue must be French, to ensure that they understand the questions asked in writing.

Control group:

- Children of the parents surveyed who do not present any medical, school or family developmental particularities.

Clinical group

- Children of the parents interviewed who present warning signs of CVI reported by a multidisciplinary team specialized in visual impairment.

Exclusion Criteria:

* no specific criteria (see inclusion criteria)

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In order to evaluate the relevance of this questionnaire, it will be proposed to parents whose children (aged 3 to 12) do not present any particular developmental difficulties, and to parents whose children (aged 3 to 12) appear to present signs of neurovisual disorders.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
typical behaviors of CVI | Through study completion, an average of 14 months
  The scores obtained represent a difficulty, an absence of mastery of a skill. Thus, a high score means that the child has some visual difficulties, while a low score means that the child has no difficulties.

CONTACTS AND LOCATIONS:
Locations (1):
- 10 place cardinal Mercier, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No